CLINICAL TRIAL: NCT06518954
Title: Self-Perceived Causes and Triggers for Eating Disorders in Athletes.
Brief Title: Triggers of Eating Disorders in Athletes
Status: Recruiting | Type: Observational
Sponsor: Ostfold University College (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Therese Fostervold Mathisen, Associate Professor, Ostfold University College
Other Study IDs: 734444
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Eating Disorders
Keywords: athlete; sport; health; illness; mental illness; eating disorder; relative energy deficiency in sport; REDs; low energy availability; LEA; body dissatisfaction; body appearance pressure; body ideal
MeSH Terms: conditions — Feeding and Eating Disorders; Mental Disorders; Relative Energy Deficiency in Sport | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athlete with eating disorder: Athletes with/with a history of eating disorder while competing in sport
  Interventions: Other: Interview
- Athlete without eating disorder: Athletes without any history of eating disorder and originating from the same club or team as the athlete with an eating disorder
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — The athletes contributes with experience exchange through individual interviews, following a interview template

SUMMARY:
Over the past 30 years, a high prevalence of eating disorders in sports has been repeatedly documented, yet few preventive measures have been implemented. While most studies explore risk factors through quantitative means, few have investigated how athletes themselves experience the triggering elements in sports and how they perceive these triggers could be better managed. Another persistent question is why some athletes from a given sport and environment develop eating disorders while others do not. This study explore the experienced triggers reported by athletes who have struggled with eating disorders and compare them to the perspectives of athletes without eating disorders from the same environment. The study also aim to gather perceptions from both groups on how eating disorders and body dissatisfaction could be better addressed and prevented in sports.

DETAILED DESCRIPTION:
Thirty years ago a Norwegian publication explored what athletes with eating disorders have experienced as the causes to their condition. Early specialization and sports cultures with early introduction to weighing and weight adjustment, high training volume, and traumatic experiences (body comments, loss of an important coach, family events) were highlighted as key self-perceived causes. This study and findings have been regularly cited and upheld as facts in professional and research literature but have not been further explored or replicated and confirmed since. This may be part of the reason why the sports world has not fully recognized its responsibility for measures despite the prevalence of eating disorders remaining unchanged over these decades. There is a need to continue exploring why some athletes develop eating disorders while others from the same conditions do not. This can be done by building on previous research and knowledge, examining specific personal or situational factors that may constitute an additional vulnerability, and also by considering self-experiences. There is also a need to understand what athletes believe can help reduce body dissatisfaction and eating disorders. This is especially relevant when considering how both the sports world and society have changed over these 30 years. Early specialization in sports, the desire to be a talent at a young age, and the massive influence of social media are factors that may be particularly challenging risk factors. Better knowledge can be used to develop supportive guidelines for sports teams and cultures, necessary rule changes, and in the education, training, and awareness of sports coaches and support staff. Such knowledge is also crucial when the sports world itself is to design the content of a national action plan to prevent body dissatisfaction and eating disorders in sports.

ELIGIBILITY:
Inclusion Criteria:

* previous/current competitive career in sport
* cohort 1: athlete with an/with a history of an eating disorder
* cohort 2: athlete from the same club without an eating disorder

Exclusion Criteria:

* disabled athletes
* not competitive athlete (below Tier 3)

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Athletes are recruited that has a past or current eating disorder, who will also suggest control individuals from the same sports team who have not had an eating disorder and can be invited to the study. These controls will serve as a comparable reference group regarding specific sports/team culture and nuances of personal experiences.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Timing of eating disorder symptoms | August-December 2024
  Question asking about when the eating disorder first started (age, performance period and level)
Cause to development of eating disorders | August-December 2024
  Question asking about what the athlete think triggered the eating disorder. comparing responses from the athlete WITH an eating disorder to the thoughts of the athlete without an eating disorder.
Knowledge on the eating disorder | August-December 2024
  Did the others in the team know about the eating disorder experienced by one of the athletes What did they observe, how did they respond or think about it, how did it affect the suffering athlete if she/he knew the others knew/did not knew.
Preventive measures | August-December 2024
  Question on what can be done to prevent eating disorders in sport. How can we better prevent eating disorders in sport; what needs to be done, what must be changed.

SECONDARY OUTCOMES:
Background variable, current symptoms of eating disorder | August-December 2024
  Eating disorder Examination Questionnaire (EDE-Q) by Prof. Fairburn. A validated questionnaire to measure symptom severity of eating disorders.
Background variable, family history | August-December 2024
  Have others in the family been diagnosed with an eating disorder (genetics), have others in the family competed in sport (environmental factors)
Background variable, other interests and identity | August-December 2024
  Have you had interests that you have invested time in, other than sport?

CONTACTS AND LOCATIONS:
Overall Officials: Therese F Mathisen, PhD, Principal Investigator — Associate Professor
Locations (2):
- Norway (2):
  - Østfold University College, Fredrikstad
  - Norwegian School of Sport Sciences, Oslo

IPD SHARING:
Plan to Share IPD: No
Interviews will not be shared with others

REFERENCES:
- [Background] Sundgot-Borgen J. Prevalence of eating disorders in elite female athletes. Int J Sport Nutr. 1993 Mar;3(1):29-40. doi: 10.1123/ijsn.3.1.29. PMID 8499936